CLINICAL TRIAL: NCT03183518
Title: A Clinical Study to Assess the Photosensitisation and Photoallergy Potential of a Cosmetic Facial Product in Healthy Subjects
Brief Title: To Assess the Photosensitisation and Photoallergy Potential of a Cosmetic Facial Product in Healthy Participants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 207587
Record Dates: First submitted 2017-05-17; First posted 2017-06-12 (Actual); Results first posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2018-06

CONDITIONS: Skin Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Product (Experimental): All the participants will have the test product applied to the appropriate test sites by trained study staff. The test site will be designated on above the waist between the left scapula and the spinal mid-line.
  Interventions: Other: Facial micellar cleanser
- Reference product (Other): All the participants will have the reference product applied to the appropriate test sites by trained study staff. The test site will be designated on above the waist between the left scapula and the spinal mid-line.
  Interventions: Other: Saline Solution: Sodium Chloride (NaCl; 0.9%)

INTERVENTIONS:
Other: Facial micellar cleanser — Each participant will have the test product applied topically via semi occlusive patch, on-site by a technician.
  Arms: Test Product
Other: Saline Solution: Sodium Chloride (NaCl; 0.9%) — Each participant will have the reference product applied topically via semi occlusive patch, on-site by a technician.
  Arms: Reference product

SUMMARY:
To evaluate the skin irritation and sensitization potential of a cosmetic facial product, under exaggerated conditions of use with controlled product application and under supervision of a dermatologist.

DETAILED DESCRIPTION:
In this three-phase phototoxicity-photosensitisation (PT-PA) study, the test material and a positive control are applied under a semi-occlusive patch to the upper back of each subject. The first phase of the study is an Induction Phase; a controlled amount of each product is applied under a semi-occlusive patch. The patch will remain on the skin for 24 (±2) hours during this phase. Following patch removal the patch site will be exposed to ultraviolet - A (UVA) radiation and re-assessed 24 hours later prior to re-application of another semi-occlusive patch (with both the products) to the same site. The Induction phase will last 3 weeks. After a subject completes the Induction Phase they will enter a Rest Phase of 2 weeks duration, during which no patches will be applied. After the Rest Phase, subjects will return to the clinical site for the Challenge Phase. In the Challenge phase two test patches will be applied to virgin skin areas on each subjects' upper back for 24 hours. Following removal of both patches, one of the Challenge patch test sites will be exposed to UVA radiation. Both Challenge patch test sites will be assessed up until 72 (±2) hours later.

ELIGIBILITY:
Inclusion Criteria

* Demonstrates understanding of the study procedures, restrictions and willingness to participate as evidenced by voluntary written informed consent and has received a signed and dated copy of the informed consent form.
* Aged between 18 and 65 years inclusive.
* Good general and mental health with, in the opinion of the investigator or medically qualified designee no clinically significant and relevant abnormalities in medical history or upon physical examination.
* Healthy, intact skin at the proposed application site; dorsum (scapular region).
* Clinical assessment for eligibility (at Visit 1 and Visit 2 - if not combined) by a dermatologist to ensure subject is free of clinically relevant dermatological conditions.
* Fitzpatrick phototype II to IV.
* Agreement to comply with the procedures and requirements of the study and to attend the scheduled assessment visits.

Exclusion Criteria

* Women who are known to be pregnant or who are intending to become pregnant over the duration of the study.
* Women who are breast-feeding.
* Any history of significant dermatological diseases or conditions or medical conditions known to alter skin appearance or physiologic response (e.g. diabetes) which could, in the opinion of the Investigator, preclude topical application of the investigational products and/or interfere with the evaluation of the test site reaction.
* Presence of open sores, pimples, or cysts at the application site.
* Active dermatosis (local or disseminated) that might interfere with the results of the study.
* Considered immune compromised.
* History of diseases aggravated or triggered by ultraviolet radiation.
* Participants with dermatographism.
* Currently using any medication which in the opinion of the investigator, may affect the evaluation of the study product, or place the subject at undue risk.
* Use of the following topical or systemic medications: immunosuppressants, antihistamines, non-hormonal anti-inflammatory drugs, and corticosteroids up to 2 weeks before screening visit.
* Oral or topical treatment with vitamin A acid and/or its derivatives up to 1 month before the screening visit.
* Intention of being vaccinated during the study period or has been vaccinated within 3 weeks of the screening visit.
* Currently receiving allergy injections, or received an allergy injection within 7 days prior to Visit 1, or expects to begin injections during study participation.
* Previous history of atopy, allergic reactions, irritation or intense discomfort feelings to topical-use products, cosmetics or medication.
* Study subjects with a history of allergy to the study material/product, hypoallergenic tape, or to the cotton patches.
* History of sensitisation in a previous patch study.
* History of abnormal reaction to sun exposure.
* Participation in another clinical study (including cosmetic studies) or receipt of an investigational drug within 30 days of the screening visit.
* Previous participation in this study.
* Recent history (within the last 5 years) of alcohol or other substance abuse.
* Intense sunlight exposure or sun tanning sessions up to 30 days before the Screening evaluation.
* Intention of bathing (in the sea or pool), sauna, water sports, or activities that lead to intense sweating.
* Any Subject who, in the judgment of the Investigator, should not participate in the study.
* Any skin marks on the test site that might interfere with the evaluation of possible skin reactions (e.g. pigmentation disorders, vascular malformations, scars, tattoos, excessive hair, numerous freckles).
* Prisoner or involuntary incarcerated subject.
* Subject from an indigenous tribe.
* An employee of the sponsor or the study site or members of their immediate family.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-03-27 (Actual); Primary Completion 2017-05-19 (Actual); Study Completion 2017-05-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Valinhos, Brazil

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants were enrolled at one center in Brazil.
Pre-assignment Details: A total of 49 participants were screened, out of which 1 participant did not meet study criteria. Remaining 48 participants were enrolled in the study, out of which 12 participants withdrew their consent before randomization.
Groups:
- All Participants: Included all participants who were randomized to receive the study treatment. In this study, the test product (cosmetic facial cleanser) and the negative control (saline solution) were randomly assigned and dispensed to 2 separated cells within a single semi-occlusive patch that was subsequently applied to the upper back (test site).
Period: Overall Study
Arm/Group | All Participants
Started | 36
Test Product (All participants received both the study treatments in single semi-occlusive patch) | 36
Negative Control (All participants received both the study treatments in single semi-occlusive patch) | 36
Completed | 33
Not Completed | 3
Not completed — Other (Not specified) | 2
Not completed — Other (Withdrawal of consent) | 1

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Baseline population includes safety population (N=36). The Safety population included all participants who received any study product.
Arm/Group | All Participants
Number analyzed (Participants) | 36
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.6 (11.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 35
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Combined Skin Irritation (Dermal Response) and Superficial Irritation (Other Effects) Scores at Induction Phase at Day 2
Description: A trained assessor assessed all patch sites. The following scores were used to express the response observed at the time of examination: 0=No evidence of irritation, 1=Minimal erythema; barely perceptible, 2=Definite erythema, readily visible; or minimal edema; or minimal papular response, 3=Erythema and papules, 4=Definite edema, 5=Erythema, edema, and papules, 6=Vesicular eruption, 7=Strong reaction spreading beyond test site. Other features indicative irritation (Superficial irritation) scores were: Grade A/Score 0=Slight glazed appearance, Grade B/Score 1=Marked glazing, Grade C/Score 2=Glazing with peeling and cracking, Grade F/Score 3=Glazing with fissures, Grade G/Score 3=Film of dried serous exudate covering all or portion of the patch, Grade H/Score 3=Small petechial erosions and/or scabs. Superficial irritation scores were only provided if there was a dermal response score >0. Full range was 0-10. Lower score indicates better tolerability.
Time Frame: At Day 2
Population: The Intent to treat (ITT, N=36) population included all participants who were randomized into the study and have skin irritation scores from at least one of the test sites available.
Measure: Mean (Standard Deviation); unit: Score on scale
Groups:
- Test Product: This arm included data from all the test sites were test product was applied.
- Negative Control: This arm included data from all the test sites were negative control was applied.
Arm/Group | Test Product | Negative Control
Number analyzed (Participants) | 36 | 36
Score on scale | 0 (0) | 0 (0)

2. Primary Outcome: Combined Skin Irritation (Dermal Response) and Superficial Irritation (Other Effects) Scores at Induction Phase at Day 4
Description: as for outcome 1
Time Frame: At Day 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Test Product | Negative Control
Number analyzed (Participants) | 36 | 36
Score on scale | 0 (0) | 0 (0)

3. Primary Outcome: Combined Skin Irritation (Dermal Response) and Superficial Irritation (Other Effects) Scores at Induction Phase at Day 5
Description: as for outcome 1
Time Frame: At Day 5
Population: The ITT (N=36) population included all participants who were randomized into the study and have skin irritation scores from at least one of the test sites available.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Test Product | Negative Control
Number analyzed (Participants) | 36 | 36
Score on scale | 0 (0) | 0 (0)

4. Primary Outcome: Combined Skin Irritation (Dermal Response) and Superficial Irritation (Other Effects) Scores at Induction Phase at Day 8
Description: as for outcome 1
Time Frame: At Day 8
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Test Product | Negative Control
Number analyzed (Participants) | 36 | 36
Score on scale | 0 (0) | 0 (0)

5. Primary Outcome: Combined Skin Irritation (Dermal Response) and Superficial Irritation (Other Effects) Scores at Induction Phase at Day 9
Description: as for outcome 1
Time Frame: At Day 9
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Test Product | Negative Control
Number analyzed (Participants) | 36 | 36
Score on scale | 0 (0) | 0 (0)

6. Primary Outcome: Combined Skin Irritation (Dermal Response) and Superficial Irritation (Other Effects) Scores at Induction Phase at Day 11
Description: as for outcome 1
Time Frame: At Day 11
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Test Product | Negative Control
Number analyzed (Participants) | 36 | 36
Score on scale | 0 (0) | 0 (0)

7. Primary Outcome: Combined Skin Irritation (Dermal Response) and Superficial Irritation (Other Effects) Scores at Induction Phase at Day 12
Description: as for outcome 1
Time Frame: At Day 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Test Product | Negative Control
Number analyzed (Participants) | 36 | 36
Score on scale | 0 (0) | 0 (0)

8. Primary Outcome: Combined Skin Irritation (Dermal Response) and Superficial Irritation (Other Effects) Scores at Induction Phase at Day 15
Description: as for outcome 1
Time Frame: At Day 15
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Test Product | Negative Control
Number analyzed (Participants) | 36 | 36
Score on scale | 0 (0) | 0 (0)

9. Primary Outcome: Combined Skin Irritation (Dermal Response) and Superficial Irritation (Other Effects) Scores at Induction Phase at Day 16
Description: as for outcome 1
Time Frame: At Day 16
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Test Product | Negative Control
Number analyzed (Participants) | 36 | 36
Score on scale | 0 (0) | 0 (0)

10. Primary Outcome: Combined Skin Irritation (Dermal Response) and Superficial Irritation (Other Effects) Scores at Induction Phase at Day 18
Description: as for outcome 1
Time Frame: At Day 18
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Test Product | Negative Control
Number analyzed (Participants) | 36 | 36
Score on scale | 0 (0) | 0 (0)

11. Primary Outcome: Combined Skin Irritation (Dermal Response) and Superficial Irritation (Other Effects) Scores at Induction Phase at Day 19
Description: as for outcome 1
Time Frame: At Day 19
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Test Product | Negative Control
Number analyzed (Participants) | 36 | 36
Score on scale | 0 (0) | 0 (0)

12. Primary Outcome: Combined Skin Irritation (Dermal Response) and Superficial Irritation (Other Effects) Scores at Challenge Phase At Week 6 (After 30 Minutes [Maximum 1 Hour], Post Patch Removal)
Description: as for outcome 1
Time Frame: At Week 6 (after 30 minutes [maximum 1 hour], post patch removal)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Test Product | Negative Control
Number analyzed (Participants) | 36 | 36
Score on scale | 0 (0) | 0 (0)

13. Primary Outcome: Combined Skin Irritation (Dermal Response) and Superficial Irritation (Other Effects) Scores at Challenge Phase At Week 6 24 (±2) Hours Post Patch Removal
Description: as for outcome 1
Time Frame: At Week 6 24 (±2) hours post patch removal
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Test Product | Negative Control
Number analyzed (Participants) | 36 | 36
Score on scale | 0 (0) | 0 (0)

14. Primary Outcome: Combined Skin Irritation (Dermal Response) and Superficial Irritation (Other Effects) Scores at Challenge Phase at Week 6 48 (±2) Hours, Post Patch Removal
Description: as for outcome 1
Time Frame: At Week 6, 48 (±2) hours, post patch removal
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Test Product | Negative Control
Number analyzed (Participants) | 36 | 36
Score on scale | 0 (0) | 0 (0)

ADVERSE EVENTS:
Time Frame: Approximately 45 days
Groups:
- All Participants: The safety population (N=36). The Safety population included all participants who received any study product.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/36
Serious Adverse Events (participants affected / at risk) | 0/36
Other Adverse Events (participants affected / at risk) | 2/36
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=36)
INFLUENZA (Infections and infestations) | 1
RHINITIS (Infections and infestations) | 1
MYALGIA (Musculoskeletal and connective tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-03-24): https://cdn.clinicaltrials.gov/large-docs/18/NCT03183518/Prot_000.pdf
  • Statistical Analysis Plan (2017-05-11): https://cdn.clinicaltrials.gov/large-docs/18/NCT03183518/SAP_001.pdf